CLINICAL TRIAL: NCT01633801
Title: Use of High Flow Ventilation in Pediatric Cardiac Surgical Patients
Brief Title: Use of High Flows in Pediatric Cardiac Surgical Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Francesca Giovanna Iodice, Doctor in Medicine, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BambinoGHRI
Record Dates: First submitted 2012-06-02; First posted 2012-07-04 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Oxygen Inhalation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High flows (Other)
  Interventions: Device: Use of high flows versus oxygen therapy; Device: oxygen therapy
- oxygen therapy (Other)
  Interventions: Device: oxygen therapy

INTERVENTIONS:
Device: Use of high flows versus oxygen therapy — Once extubation has taken place the child will be placed either on traditional oxygen therapy or high flow nasal cannulae according to randomization.
  Other Names: high flow nasal cannulae; (via Neonatal Nasal Cannula- Fisher & Paykel)
  Arms: High flows
Device: oxygen therapy — Once extubation has taken place the child will be placed either on traditional oxygen therapy or high flow nasal cannulae according to randomization.
  Other Names: traditional nasal cannulae

SUMMARY:
Humidified high flow nasal prong oxygen therapy is a method for providing oxygen and CPAP. The delivery of high flows decreases dilution of the inhaled oxygen and, by matching patient's peak flow, allows accurate delivery of the set FiO2 throughout the whole inspiratory phase. In addition, a flow-dependent effect of continuous positive airway pressure, possibly due to an air entrainment mechanism, has been documented in healthy volunteers and in patients with COPD.

The investigators working hypothesis is that the use of post-extubation CPAP delivered via nasal cannulae in infants less than 18 months, post-bypass surgery will have better PaCO2 values than infants extubated on to oxygen therapy.

DETAILED DESCRIPTION:
After CICU admission, infants with no bleeding, normothermic and hemodynamically stable will be switched from PRVC to SIMV+PSV (10-15cmH20) which should be maintained for 4 hours. An arterial gas analysis will be performed after 20 minutes. Infants with normal gas-exchange are gradually weaned from mechanical ventilation At each weaning step an arterial hemogasanalysis is performed after 20 minutes, to assess if the decreased ventilatory support is tolerated. Increased work of breathing and respiratory acidosis (ph< 7.3 or pCO2 > 60 mmHg) are considered criteria to withhold the weaning process. After a 4 hour period on SIMV+PSV the child should be switched to PSV for 30 minutes and then extubated. The following extubation criteria should be reached:

* Satisfactory blood gases with PCO2 under 45mmHg, pH greater than 7.30.
* Fractional inspired oxygen concentration of 65% and or less than the baseline value
* Adequate respiratory frequency according to age without dyspnea

At this point criteria for extubation are reached. Once extubation has taken place the child will be placed either on traditional oxygen therapy or high flow nasal cannulae according to randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age: 0-18 months
* Mechanical Ventilation via an endotracheal tube
* Elective surgery
* Post-bypass procedure
* Rachs 2 and above

Exclusion Criteria:

* Presence of major congenital malformations
* Presence of neuromuscular disease
* Presence of non drained pneumothorax
* Absent respiratory drive or recurrent apneas
* Hemodynamic instability
* Glasgow coma score (GCS) less than 8
* ECG with evidence of ischaemia or arrhythmias
* Active bleeding

Ages: 1 Day to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2012-08; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The primary aim of this study is to show an improvement of the average levels of postextubation PaCO2 in infants less than 18 months of age and post-bypass surgery | Final outcome measure is assessed when 80 patients have been recruited.Outcome measure is assessed at the end of 48 hours postextubation and when the patient is discharged from the ICU.

SECONDARY OUTCOMES:
The secondary aim is to verify the reintubation rate between the two groups. | Final outcome measure is assessed when 80 patients have been recruited.Outcome measure is assessed at the end of 48 hours postextubation and when the patient is discharged from the ICU.
  Other points that will be evaluated are: the improvement of X-ray findings, the length of ICU stay and the development of complications such as nasal ulcers and gastric distension.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Iodice, MD, Principal Investigator — Ospedale Bambino Gesu'
Locations (2):
- Italy (2):
  - Francesca Iodice, Rome, Italy
  - Ospedale Bambino Gesu, Rome

REFERENCES:
- [Derived] Testa G, Iodice F, Ricci Z, Vitale V, De Razza F, Haiberger R, Iacoella C, Conti G, Cogo P. Comparative evaluation of high-flow nasal cannula and conventional oxygen therapy in paediatric cardiac surgical patients: a randomized controlled trial. Interact Cardiovasc Thorac Surg. 2014 Sep;19(3):456-61. doi: 10.1093/icvts/ivu171. Epub 2014 Jun 8. PMID 24912486